CLINICAL TRIAL: NCT03847597
Title: Histological and Imaging Assessment of the Structural Characteristics of the Femoro-popliteal Arterial Segment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7168
Record Dates: First submitted 2018-12-18; First posted 2019-02-20 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-12

CONDITIONS: Chronic Limb Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Explantation of the femoro-popliteal arterial segment from the amputed limb — Explantation of the femoro-popliteal arterial segment from the amputed limb

SUMMARY:
The femoro-popliteal arterial segment is one of the most frequent locations for atherosclerosis. Its management is mainly endovascular (standard and coated-balloon angioplasty, stenting).

However, the structural features of the atherosclerotic disease in regards to patient's risk factors and past medical and surgical histories are not well studied. Furthermore, the histological analysis of the femoro-popliteal arterial segment is rare in the literature, and made difficult mostly because of the length of this segment.

There is a clinical need for better understanding of atherosclerotic lesions in this location, with as further goal, a better management of this disease.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years old
* Men and women
* Patient with chronic limb ischemia that is scheduled for transfemoral amputation in the University Hospital of Strasbourg
* Patient giving his -non-opposition to the explantation and use of the femoro-popliteal arterial segment

Exclusion criteria:

* Refusal to give his consent
* Impossibility to give clear information to the patient
* Pregnant and breastfeeding women
* Patient under administrative protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic limb ischemia that are scheduled for transfemoral amputation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the arterial structure in micro-CT. | 3 years
  study precisely the pathological structure of the femoro-popliteal arterial segment in AOMI, both in imaging and histologically.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil CHAKFE, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided